CLINICAL TRIAL: NCT06663553
Title: Protocol for a Comparative Study of the Efficacy of Transumbilical Laparoendoscopic Single-site Surgery (TU-LESS) and Transvaginal Natural Orifice Transluminal Endoscopic Surgery (vNOTES) in Hysterectomy Performed on Patients With Enlarged Uterus: A Prospective Single-blinded, Randomized Clinical Trial
Brief Title: Comparing the Efficacy of TU-LESS and vNOTES for Hysterectomy of Enlarged Uterus
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West China Second University Hospital (Other)
Responsible Party: Principal Investigator, Hongyu Jin, lecturer and gynecological surgeon, West China Second University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020079JHY
Record Dates: First submitted 2024-10-19; First posted 2024-10-29 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-08

CONDITIONS: Enlarged Uterus; Adenomyosis; Uterine Fibroids (UF)
MeSH Terms: conditions — Adenomyosis; Leiomyoma

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients will remain blinded to their surgical methods in 24 hours following the operation. To achieve this, we will apply wound pads to each patient's abdomen as the wounds typically seen in tradi tional laparoscopy procedures, no matter whether actual wounds exist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TU-LESS for hysterectomy (Active Comparator): Patients diagnosed with enlarged uteri following a bimanual examination, with confirmation of the size and nature of the enlargement through imaging techniques such as ultrasound or magnetic resonance imaging (MRI).
  Interventions: Procedure: TU-LESS
- vNOTES for hysterectomy (Experimental): Patients diagnosed with enlarged uteri following a bimanual examination, with confirmation of the size and nature of the enlargement through imaging techniques such as ultrasound or magnetic resonance imaging (MRI).
  Interventions: Procedure: vNOTES

INTERVENTIONS:
Procedure: TU-LESS — patients in TU-LESS group will receive transumbilical laparoendoscopic single-site surgery (TU-LESS) for hysterectomy
  Arms: TU-LESS for hysterectomy
Procedure: vNOTES — patients in vNOTES group will receive transvaginal natural orifice transluminal endoscopic surgery (TU-LESS) for hysterectomy
  Arms: vNOTES for hysterectomy

SUMMARY:
Enlarged uterus is frequently encountered in clinical practice, and its incidence due to conditions such as adenomyosis, uterine fibroids, and other gynecological disorders has steadily increased over the years statistically. For example, greater healthcare awareness has led to more frequent early diagnoses of these conditions, contributing to the observed rise in incidence. Additionally, increasing life expectancy results in more women reaching the perimenopausal and postmenopausal stages, during which conditions like uterine fibroids and adenomyosis become more prevalent. For these women, hysterectomy (removal of the entire uterus) is often the recommended option of treatment.

With advances in surgical techniques over recent decades, there has been a notable shift from traditional open abdominal surgeries to minimally invasive approaches. Laparoscopic surgery has been widely adopted, significantly reducing the size and number of incisions required, thereby promoting faster recovery, minimizing postoperative pain, and reducing the risk of complications.

However, conventional multi-port laparoscopic hysterectomy still presents certain challenges, such as large uterus extraction following resection, and concerns about healing of incisions. In contrast, innovative techniques like Transumbilical Laparoendoscopic Single-Site Surgery(TU-LESS) and Transvaginal Natural Orifice Transluminal Endoscopic Surgery(vNOTES) both take advantage of natural anatomical openings to achieve minimal or no visible scarring. Studies demonstrate that these techniques provide superior outcomes in terms of reduced pain, faster recovery, and quicker return to daily activities compared to traditional multi-port laparoscopic approaches.

Yet a direct comparison of the efficacy of these two methods in real-world, particularly for enlarged uterus, remains inconclusive. Thus this study aims to evaluate and compare the outcomes of these two techniques in patients with enlarged uteri. Participants will be randomly assigned to receive one of the two surgical approaches, ensuring an unbiased comparison of the efficacy of the procedures in terms of healing status and recovery time.

DETAILED DESCRIPTION:
Enlarged uterus, mainly caused by adenomyosis, is often associated with symptoms like compression of intestines and urethra(presenting as constipation, urinary frequency, and urgency), dysmenorrhea, menstrual irregularity, and anemia due to menorrhagia. A hysterectomy (removal of the uterus) is often recommended, especially in cases where conservative management like medical treatment fails.

Among all the methods of hysterectomy, TU-LESS and vNOTES are noted for minimized invasiveness and fast recovery. As vNOTES is performed through the vagina and TU-LESS involves a single incision through the umbilicus, they both utilize natural anatomical openings, resulting in minimal to no visible scarring.

ELIGIBILITY:
Inclusion Criteria:

* Eligible women aged 18-70 years.
* Women with indications for enlarged uterine volumes who are planning to under go total hysterectomy. Uterine size should exceed that of a 3-month pregnancy (uterine weight ≥ 280 g).
* Patients are willing to be randomly assigned to undergo any of both approaches.
* Patients who are willing to sign the informed consent form.

Exclusion Criteria:

* Individuals who are virgins or have vaginal stenosis.
* Patients requiring concurrent surgical intervention for conditions such as ovarian cysts or lesions of the vulva, vagina, appendix, etc.
* presence of uterus exceeding approximately 20 gestational weeks in size (about 900-1000g), which is beyond the limitations of a single-site laparoscopic approach due to concerns regarding technical feasibility and safety
* Presence of malignancy or strong suspicion of malignancy that may alter the planned surgical approach.
* History of two or more pelvic surgeries or suspected severe pelvic adhesions (rectovaginal examination suggesting rectovaginal endometriosis or limited uterine mobility).
* History of peritoneal dialysis, pelvic radiation therapy and pelvic tuberculosis treated with laparoscopic surgery.
* Patients with prolapse or pelvic inflammation.
* Diabetes mellitus with poor blood glucose control.
* Body mass index greater than 30 kg/m².

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Enlarged uterine volumes occur only to female population
Enrollment: 210 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
postoperative liquid diet | within 24 hours postoperatively
  the proportion of patients able to consume a liquid diet post-surgery
passing flatus | within 24 hours postoperatively
  the proportion of patients able to pass flatus
self-urination after catheter removal | within 24 hours postoperatively
  The proportion of patients regaining the ability to urinate without assistance after catheter removal
ambulation | within 24 hours postoperatively
  The proportion of patients regaining mobility after catheter removal
hospital stay | within 2 days postoperatively
  The percentage of patients discharged within 2 days after surgery
examination of pelvic fuction | within 2 days postoperatively
  The assessment of pelvic floor function involves evaluating Stress Urinary Incontinence (SUI), Pelvic Organ Prolapse (POP) and Sexual Dysfunction.
  The PISQ-IR (Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire) is a validated tool specifically designed to evaluate sexual function in the context of pelvic floor. It is a tool that measures sexual function specifically for women affected by pelvic floor disorders, such as urinary incontinence and pelvic organ prolapse.

SECONDARY OUTCOMES:
Postoperative pain | at 12 hours and 24 hours postoperatively
  It is measured by the VAS score. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').
The duration of operation | during operation
  It will be measured in min utes, starting from the initiation of the skin (or vag inal) incision and concluding upon the completion of the skin (or vaginal) suturing. If a frozen biopsy is needed during the operation, the increased time for the frozen biopsy should be subtracted. However, pa tients for whom the surgical method is changed due to the result of the frozen biopsy should be excluded.
amount of bleeding | during operation
Intraoperative complications and postoperative complications | within 3 months
  We use the Clavien-Dindo classification to rank a complication in an objective and reproducible manner.
  It consists of 7 grades (I, II, IIIa, IIIb, IVa, IVb and V). The introduction of the subclasses a and b allows a contraction of the classification into 5 grades (I, II, III, IV and V) depending on the size of the population observed or the of the focus of a study.
abdominal scars assessment | both at 3 and 6 months after surgery
  The Patient and Observer Scar Assessment Scale (POSAS) will be used. It consists of two separate scales: the Patient Scale and the Observer Scale and measures scar quality (i.e. how the scar looks and feels) from both perspectives.
  The observer scores six items: vascularization, pigmentation, thickness, surface roughness, pliability, and surface area. The patient scores six items: pain, pruritus, color, thickness, relief, and pliability.
  All included items are scored on the same polytomous 10-point scale, in which a score of 1 is given when the scar characteristic is akin to 'normal skin' and a score of 10 reflects the 'worst imaginable scar'. All items are summed to give a total scar score, and therefore, a higher score represents a poorer scar quality.
the total dosage of analgesics taken | during the first 24 hours following surgery
  also categorized by analgesic type
The Female Sexual Function Index(FSFI) | both at baseline and 6 months after surgery
  Using either a paper sheet or online questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- West China Second University Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Background] Benassi L, Rossi T, Kaihura CT, Ricci L, Bedocchi L, Galanti B, Vadora E. Abdominal or vaginal hysterectomy for enlarged uteri: a randomized clinical trial. Am J Obstet Gynecol. 2002 Dec;187(6):1561-5. doi: 10.1067/mob.2002.127596. PMID 12501064
- [Background] Zhang W, Deng L, Yang F, Liu J, Chen S, You X, Gou J, Zi D, Li Y, Qi X, Wang Y, Zheng Y. Comparing the efficacy and safety of three surgical approaches for total hysterectomy (TSATH): protocol for a multicentre, single-blind, parallel-group, randomised controlled trial. BMJ Open. 2024 Jan 10;14(1):e074478. doi: 10.1136/bmjopen-2023-074478. PMID 38199630
- [Derived] Chen X, Zhang M, Gao M, Wu Y, He Y, Liu J, Cui H, Jin H. Protocol for a study comparing the efficacy of hysterectomy in patients with enlarged uterus via TU-LESS and vNOTES: a single-blind, prospective randomised clinical trial. BMJ Open. 2025 Nov 26;15(11):e103174. doi: 10.1136/bmjopen-2025-103174. PMID 41298256